CLINICAL TRIAL: NCT02119689
Title: Vascular Reparative Mechanism by ACE2/Ang-(1-7) in Diabetes
Brief Title: Vascular Reparative Mechanism in Diabetes
Acronym: RAAS
Status: Active, not recruiting | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Maria Grant, Professor, University of Alabama at Birmingham
Other Study IDs: 1308798827; R01HL110170 (NIH)
Record Dates: First submitted 2014-04-14; First posted 2014-04-22 (Estimated); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Diabetic Retinopathy
Keywords: Diabetes; Retinopathy
MeSH Terms: conditions — Diabetic Retinopathy; Diabetes Mellitus; Retinal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Diabetic Patients: Mild, Moderate and Severe Retinopathy
  Interventions: Other: Diabetic Patients
- Healthy Controls: Age and sex matched Healthy Controls
  Interventions: Other: Healthy Controls

INTERVENTIONS:
Other: Diabetic Patients — measuring CD34 cell function in relation to diabetic retinopathy status
  Groups: Diabetic Patients
Other: Healthy Controls — measuring CD34 cell function
  Groups: Healthy Controls

SUMMARY:
The purpose of this research study is to study blood stem cells in diabetic patients and normal patients. We would like to better understand if these cells, called endothelial precursor cells (EPCs), are not working as expected in people with diabetes. We would like to see if the function of these cells can predict the development of diabetic retinopathy.

Diabetic retinopathy is an eye disease associated with diabetes in which the cells of the retina are damaged. It can cause blurred vision, vision loss, blindness or possible bleeding in the retina. Even with current treatments, the quality of life for people with diabetic retinopathy is much reduced.

ELIGIBILITY:
Inclusion Criteria:

* Men or women 18 years or older
* 39 type 1 or type 2 diabetic patients
* 13 with mild retinopathy
* 13 with moderate retinopathy
* 13 with severe, nonproliferative retinopathy
* 39 age and sex matched healthy controls

Exclusion Criteria:

* Current pregnancy as evidence by a urine pregnancy test as the blood from a pregnant female will influence the results of the laboratory tests

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Ophthalmology and Primary Care Clinics
Sampling Method: Probability Sample
Enrollment: 78 (Estimated)
Dates: Start 2011-10-30 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The ACE/ACE2 ratio within EPC's | up to 216 weeks
  Peripheral blood of 150cc, approximately 8-10 tablespoons will be collected from a vein in the arm of both diabetic and healthy control patients.

SECONDARY OUTCOMES:
The balance of the RAS (renin-angiotensin system) within EPCs | up to 216 weeks
  The Endo-PAT2000 will be used to obtain this measurement. This is a 15-minute office-based test where a blood-pressure cuff is placed around the arm, inflated and measurements are obtained from a small fingertip monitor

OTHER OUTCOMES:
Photography findings | up to 216 weeks
  The findings from eye photographs will be collected and evaluated from both the diabetic patients and the heallthy control patients. This will be done at either the patient's yearly visit or at their 6 week follow-up visit.
Fluorescein angiogram findings | up to 216 weeks
  The findings from eye photographs will be collected and evaluated from both the diabetic patients and the heallthy control patients. This will be done at either the patient's yearly visit or at their 6 week follow-up visit.

CONTACTS AND LOCATIONS:
Overall Officials: Maria B Grant, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama, Birmingham, Alabama, United States